CLINICAL TRIAL: NCT06532331
Title: A PhaseⅠStudy to Examine Tolerability and Safety of ONO-7475 in Combination With ONO-4538 and Gemcitabine Plus Nab-paclitaxel (GnP), the Standard of Care, and Safety of ONO-7475 in Combination With GnP in Patients With Metastatic Pancreatic Cancer as First-line Treatment
Brief Title: A PhaseⅠStudy of ONO-7475 in Combination With ONO-4538 and Gemcitabine Plus Nab-paclitaxel (GnP), the Standard of Care, and ONO-7475 in Combination With GnP in Patients With Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONO-7475-04
Record Dates: First submitted 2024-07-28; First posted 2024-08-01 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-7475+GnP (Experimental)
  Interventions: Drug: ONO-7475; Drug: Nab-paclitaxel; Drug: Gemcitabine
- ONO-7475＋ONO-4538＋GnP (Experimental)
  Interventions: Drug: ONO-7475; Drug: ONO-4538; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: ONO-7475 — Specified dose on specified days
Drug: ONO-4538 — Specified dose on specified days
  Other Names: Nivolumab
  Arms: ONO-7475＋ONO-4538＋GnP
Drug: Nab-paclitaxel — Specified dose on specified days
Drug: Gemcitabine — Specified dose on specified days

SUMMARY:
This study is PhaseⅠstudy to examine tolerability and safety of ONO-7475 in combination with ONO-4538 and gemcitabine plus nab-paclitaxel (GnP), the standard of care, and safety of ONO-7475 in combination with GnP in patients with metastatic pancreatic cancer as first-line treatment

ELIGIBILITY:
Inclusion Criteria:

1. Patient with metastatic pancreatic cancer
2. Patients have an ECOG performance status of 0 to 1
3. Patients with a life expectancy of at least 6 months

Exclusion Criteria:

1. Patients are unable to swallow oral medications
2. Patients with severe complication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | 28 days
Adverse event (AE) | Up to 28 days after the last dose

SECONDARY OUTCOMES:
Pharmacokinetics (Plasma concentration of ONO-7475) | Up to Cycle16
Pharmacokinetics (Plasma concentration of ONO-4538) | Through study completion, an average of 6 months
Anti-ONO-4538 antibody | Through study completion, an average of 6 months
Objective Response Rate (ORR) | Through study completion, an average of 6 months
Disease Control Rate (DCR) | Through study completion, an average of 6 months
Overall Survival (OS) | Through study completion, an average of 1 year
Progression-Free Survival (PFS) | Through study completion, an average of 6 months
Duration of Response (DOR) | Through study completion, an average of 6 months
Time to Response (TTR) | Through study completion, an average of 6 months
Best Overall Response (BOR) | Through study completion, an average of 6 months
Percent change in the sum diameters of the target lesions | Through study completion, an average of 6 months
Maximum percent change in the sum diameters of the target lesions | Through study completion, an average of 6 months
CEA | Through study completion, an average of 6 months
CA19-9 | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (9):
- Japan (9):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Osaka International Cancer Institute, Osaka, Osaka
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Juntendo University Hpspital, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR, Koto-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No